CLINICAL TRIAL: NCT02351232
Title: The Lira Pump Trial. The Effects of Liraglutide in Patients With Insulin Pump Treated Type 1 Diabetes: A Randomized Placebo-Controlled Trial
Brief Title: The Lira Pump Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Signe Schmidt, MD, PhD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LPT2015; 2014-002285-76 (EudraCT Number)
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2016-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Liraglutide; daily subcutaneous injection; 1.8 mg; 6 months
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Placebo; daily subcutaneous injection; 1.8 mg; 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide
  Other Names: Victoza
  Arms: Intervention
Drug: Placebo
  Arms: Placebo

SUMMARY:
A randomized placebo-controlled clinical trial investigating the effects of Liraglutide as an add-on to intensive insulin therapy in overweight insulin pump treated type 1 diabetes patients in suboptimal glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes ≥ 1 year
* BMI > 25 kg/m2
* Insulin pump ≥ 1 year
* HbA1c > 58 mmol/mol
* Use of carbohydrate counting and the insulin pump bolus calculator

Exclusion Criteria:

* Gastroparesis
* Impaired renal function (eGFR < 60 ml/min/1.73m2)
* Liver disease with ALAT > 2.5 times the upper limit of the reference interval
* Acute or chronic pancreatitis or history of chronic pancreatitis or idiopathic acute pancreatitis
* Inflammatory bowel disease
* History of cancer (except basal cell skin cancer) which in the investigators opinion could interfere with the results of the trial, or cancer during the past 5 years
* Thyroid adenoma
* Subjects with personal or family history of MTC or MEN2
* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period or within 30 days prior to study start
* Known or suspected alcohol or drug abuse
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the patient unsuitable for study participation
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods.
* Simultaneous participation in any other clinical intervention trial
* Known or suspected hypersensitivity to Liraglutide
* Inability to understand the patient information and to give informed consent
* Acute treatment required proliferative retinopathy or maculopathy (macular oedema)
* Any Cardiac disorder which in the investigators opinion could interfere with the safety and results of the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 6 months
  Change in HbA1c from baseline to end of study (time 6 months)

SECONDARY OUTCOMES:
Change in weight | 6 months
  Change in weight from baseline to end of study (time 6 months)
Change in insulin pump settings | 6 months
  Change in insulin pump settings from baseline to 3 weeks, 3 months and 6 months
Change in glucose variability as measured by continuous glucose monitoring | 6 months
  Change in glucose variability from baseline to 3 weeks, 3 months and 6 months
Change in body composition as measured by DXA-scan | 6 months
  Change in body composition from baseline to 6 months
Change in blood pressure | 6 months
  Change in blood pressure from baseline to 6 months
Change in lipid profile (LDL, HDL, VLDL, total cholesterol, triglycerides) | 6 months
  Change in lipid profile from baseline to 6 months
Frequency of hypoglycemia (patient reported number of episodes with blood glucose <3.9 mmol/l) | 6 months
  Frequency of hypoglycemia during the 6-month study period
Change in kidney function as measured by urine albumine/creatinine ratio | 6 months
  Change in kidney function from baseline to 6 months
Number of daily blood glucose measurements | 6 months
  Number of daily blood glucose measurements during the 6-month study period
Change in diet as measured by retrospective food recording | 6 months
  Change in dietary behavior from baseline to 3 and 6 months
Change in treatment satisfaction as measured by Diabetes Treatment Satisfaction Questionnaire | 6 months
  Change in treatment satisfaction from baseline to 3 and 6 months
Change in anxiety and depression as measured by Hospital Anxiety and Depression Scale | 6 months
  Change in anxiety and depression from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Nørgaard, MD, DMSc, Principal Investigator — Hvidovre University Hospital
Locations (2):
- Denmark (2):
  - Steno Diabetes Center, Gentofte Municipality
  - Hvidovre University Hospital, Hvidovre

REFERENCES:
- [Result] Dejgaard TF, Schmidt S, Frandsen CS, Vistisen D, Madsbad S, Andersen HU, Norgaard K. Liraglutide reduces hyperglycaemia and body weight in overweight, dysregulated insulin-pump-treated patients with type 1 diabetes: The Lira Pump trial-a randomized, double-blinded, placebo-controlled trial. Diabetes Obes Metab. 2020 Apr;22(4):492-500. doi: 10.1111/dom.13911. Epub 2019 Dec 19. PMID 31696598